CLINICAL TRIAL: NCT01414712
Title: Circulating Tumor Cells in Patients Undergoing Stereotactic Body Radiotherapy for Low- and Intermediate-Risk Prostate Cancer
Brief Title: Circulating Tumor Cells in Prostate Cancer Patients
Status: Terminated | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STU 032011-212
Record Dates: First submitted 2011-05-18; First posted 2011-08-11 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2013-03

CONDITIONS: Prostate Cancer
Keywords: Low- and Intermediate-Risk Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- prostate cancer patients
  Interventions: Other: Blood Drawing

INTERVENTIONS:
Other: Blood Drawing — Blood Drawing to measure circulating tumor cells counts.
  Other Names: Blood Drawing for prostate cancer patients who undergo stereotactic body radiotherapy

SUMMARY:
The purpose of this study is to determine if a non-invasive cancer treatment, high-dose stereotactic body radiotherapy (SBRT), is associated with changes in circulating tumor cells counts in patients with low- and intermediate-risk prostate cancer.

DETAILED DESCRIPTION:
SBRT (stereotactic body radiotherapy) may decrease or actually increase CTC levels in patients with cancer, and knowledge about the effects of different therapies, including SBRT, on CTC levels will be of general interest to the oncology community. Patients will undergo blood draws at defined times as indicated below.

1. Prior to CT-simulation, but more than 2 days after digital rectal examination
2. Within 24 hours following CT simulation (an endorectal balloon is used at the time of simulation)
3. Within 24 hours following the first treatment
4. Within 24 hours following the third treatment
5. Within 1 week following the fifth treatment

ELIGIBILITY:
Inclusion Criteria:

Men who satisfy all of the following conditions will be eligible for this study:

* Willing and capable to provide informed consent
* Signed study specific informed consent form.
* PSA ≤ 20 prior to hormone therapy (if given) for patients with Gleason 2-6. For those with Gleason score of 7. PSA should be less than or equal to 15 ng/ml prior to hormonal therapy (if given). Thus, risk of pelvic lymph node involvement according to Roach formula would be under 20%.
* Gleason score ≤ 7
* Appropriate staging studies identifying as AJCC stage T1a, T1b, T1c, T2a, or T2b
* No direct evidence of regional or distant metastases after appropriate staging studies
* Histologic confirmation of cancer by biopsy
* Adenocarcinoma of the prostate
* Age ≥ 18
* Zubrod Performance Status 0-2
* Up to 9 months of previous hormonal therapy is allowed (but not required)
* AUA score must be ≤ 15 (alpha blockers allowed)
* CT or Ultrasound-based volume estimation of prostate gland ≤ 60 grams
* Agreement to use effective contraceptive methods such as condom/diaphragm and spermicidal foam, intrauterine device, or prescription birth control pills.

Exclusion Criteria:

Women are not eligible for this study. Men with one or more of the following conditions also are ineligible for this study:

* Positive lymph nodes or metastatic disease from prostate cancer
* Prior invasive malignancy unless disease free for a minimum of 3 years (carcinoma in situ of the breast, oral cavity, or cervix, or non-melanomatous skin cancer are all permissible)
* T2c, T3, or T4 tumors
* Previous pelvic radiotherapy
* Previous surgery or chemotherapy for prostate cancer
* Previous transuretheral resection of the prostate (TURP) or cryotherapy to the prostate
* Previous hormonal therapy given for more than 9 months prior to therapy
* Concomitant antineoplastic therapy (including surgery, cryotherapy, conventionally fractionated radiotherapy, and chemotherapy) while on this protocol.
* History of Crohn's Disease or Ulcerative Colitis.
* Previous significant obstructive symptoms; AUA score must be ≤ 15 (alpha blockers allowed)
* Significant psychiatric illness
* Men of reproductive potential may not participate unless they agree to use an effective contraceptive method.
* Ultrasound or CT estimate of prostate volume > 60 grams

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Low- and Intermediate-Risk Prostate Cancer wo undergo stereotactic body radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To review the level of changes in circulating tumor cells with radiation. | 2 weeks
  The investigator will review the coutns of circulating tumor cells (CTC). If there are significant changes in CTC levels with radiation, future studies will determine the prognostic significance of this information.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States